CLINICAL TRIAL: NCT06473831
Title: Creation of Side-to-Side Compression Anastomosis Using the GT Metabolic Solutions Magnet System, DI Biofragmentable (MagDI System) in Australia to Achieve Duodeno-Ileostomy Diversion in Adults With Obesity and With or Without Type 2 Diabetes Mellitus (MagDI Australia Study)
Brief Title: MagDI Australia Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GT Metabolic Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTM-009
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is an open-label multicenter study enrolling up to 30 participants at up to 3 sites in Australia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnet System, DI Biofragmentable (Experimental): GT Metabolic Solutions Magnet System, DI Biofragmentable (MagDI System)
  Interventions: Device: Magnet System, DI Biofragmentable

INTERVENTIONS:
Device: Magnet System, DI Biofragmentable — Anastomoses achieved by magnetic compression.

SUMMARY:
The objective of the MagDI Australia Study is to evaluate the feasibility / performance, safety, and initial efficacy of the MagDI System in eligible participants who are indicated for a duodeno-ileal (small bowel) side-to-side anastomosis procedure for partial intestinal diversion (e.g., one example of a small bowel clinical procedure requiring a side-to-side anastomosis).

DETAILED DESCRIPTION:
The objective of the MagDI Australia Study is to evaluate the feasibility / performance, safety, and initial efficacy of the MagDI System in eligible participants who are indicated for a duodeno-ileal (small bowel) side-to-side anastomosis procedure for partial intestinal diversion (e.g., one example of a small bowel clinical procedure requiring a side-to-side anastomosis).

The partial diversion of intestinal contents from the duodenum to the ileum via side-to-side duodeno-ileostomy is intended to facilitate weight management / loss in obese adults and improve metabolic outcomes in obese adults with and without type 2 diabetes mellitus (T2DM). Side-to-side anastomoses are currently created by sutures, staples, and anastomotic compression devices. The most common side-to-side anastomosis technique used today is stapling, requiring cutting of the intestines and staples remain behind in the body. Linear staplers are available in different sizes (e.g., 30mm, 45mm, 50mm, 60mm). A predicate for this side-to-side duodeno-ileostomy diversion procedure is the single-anastomosis duodeno-ileostomy (SADI) procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18-65 years of age, at the time of informed consent.
2. Body Mass Index (BMI) between 30-50 kg/m2
3. Meets one of the following criteria:

   1. Type 2 Diabetes Mellitus (T2DM; defined as HbA1c ≥ 6.5%) following previous sleeve gastrectomy (≥ 12 months); OR
   2. Type 2 Diabetes Mellitus (T2DM; defined as HbA1c ≥ 6.5%) without previous sleeve gastrectomy and without plan to perform a concurrent sleeve gastrectomy.
   3. Weight regain following previous sleeve gastrectomy (≥ 12 months).
4. Participant agrees to refrain from any type of additional bariatric or reconstructive surgery that would affect body weight for the duration of the study.
5. Participant has been informed of the nature of the study and agrees to its provisions, complying with study required testing, medications, follow-up visits, and has provided written informed consent.
6. Participant is indicated for, and has agreed to, a bariatric procedure involving a duodenal ileal anastomosis. The participant has also undergone the site standard of care evaluation for this type of procedure, which is expected to involve clinical assessments over a period of time by a multidisciplinary team and may include, but is not limited to, the following: screening for surgical safety, interviews to determine if the participant understands the procedure and post-operative demands, and whether the participant has the necessary social supports in place to help manage outcomes.

Exclusion Criteria:

1. Type 1 diabetes.
2. Use of injectable insulin.
3. Uncontrolled Type 2 Diabetes Mellitus (T2DM).
4. Investigator plans to perform a sleeve gastrectomy with the duodeno-ileal anastomosis procedure.
5. Uncontrolled hypertension, dyslipidemia or sleep apnea.
6. Prior intestinal, colonic or duodenal surgery (other than bariatric).
7. Prior surgery, trauma, prostheses, disease or genetic expression which prevent or contraindicate the procedure, including scarring and abnormal anatomy.
8. Refractory gastro-esophageal reflux disease (GERD).
9. Barrett's disease.
10. Helicobacter pylori positive and/or active ulcer disease.
11. Large hiatal hernia.
12. Inflammatory bowel or colonic diverticulitis disease.
13. Any anomaly precluding orogastric access by gastroscope and catheters, and manipulation techniques.
14. Any anomaly preventing / contraindicating endoscopic or laparoscopic access and procedures.
15. Implantable pacemaker or defibrillator.
16. Psychiatric disorder, except well-controlled depression with medication for > 6 months.
17. History of substance abuse.
18. Pregnant, lactating, or planning pregnancy during the clinical investigation. Note: Female participants of childbearing age must agree to use safe contraception (e.g., intrauterine devices, hormonal contraceptives: contraceptive pills, implants, transdermal patches hormonal vaginal devices, injections with prolonged release).
19. Any comorbidity or current status of participant's physiological fitness that in the surgeon's or anesthesiologist's opinion represents safety concerns that make the participant medically unfit for the procedure, including any significant congenital or acquired anomalies of the GI tract at or distal to the placement of the Magnets.
20. Unhealed ulcers, bleeding lesions, tumor, or any other lesion at target Magnet deployment site.
21. Expected need for Magnetic Resonance Imaging (MRI) within the first 2 months post-procedure.
22. Any surgical or interventional procedure (including planned and/or scheduled) within the period of 30 days prior to and 30 days following the study procedure.
23. Any stroke/TIA ≤ 6 months prior to consent.
24. Requires chronic anticoagulation therapy (except aspirin).
25. Active infections requiring antibiotic therapy, unless resolved before undergoing the study procedure.
26. Recent tobacco or nicotine product cessation ≤ 3 months prior to informed consent.
27. Known allergies to the device components (including the biofragmentable material PGLA or similar compounds) or contrast media.
28. Participants with comorbidities that are likely to result in a life expectancy of ≤ 12 months.
29. Currently participating in an investigational drug or another device study that has not reached its primary endpoint: Note: Studies requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.
30. A positive COVID-19 test prior to the study procedure in accordance with local COVID-19 protocol.
31. Presence of other anatomic or comorbid conditions, or other medical, social or psychological conditions that, in the investigator's opinion, could limit the participant's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Feasibility and performance of the side-to-side anastomosis for duodeno-ileal diversion using the MagDI System. | From date of study index procedure through 90 days
  The duodeno-ileal diversion will be considered feasible if it results in successful:
  * Placement of the Magnet System (≥ 90% alignment of magnets); and
  * Creation of a patent anastomosis confirmed radiologically, and
  * Passage of magnets without any surgical re-interventions.
  The primary endpoint will be met if the feasibility/performance is confirmed in ≥ 80% of enrolled and treated subjects.
Safety of the MagDI System | Procedure, Day 90, Day 180, Day 360
  Freedom from serious adverse events related to the study device or study device procedure requiring additional emergency surgery or re-intervention, including:
  * All-cause mortality
  * Intestinal perforation and/or peritonitis
  * Intestinal obstruction
  * Life-threatening bleeding
  * Incidence of device malfunctions

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Dr. Mark Magdy (affiliated with St. George Private Hospital), Sydney, New South Wales
  - St. John of God Health Care, Inc., Murdoch, Western Australia
  - Calvary Health Care Adelaide Limited, Adelaide
  - Upper GI Surgery, Sydney

IPD SHARING:
Plan to Share IPD: No